CLINICAL TRIAL: NCT01272648
Title: Rehabilitation and Coping of Effects After Curative Radiotherapy for Prostate
Brief Title: Rehabilitation After Radiotherapy for Prostate Cancer
Acronym: RePCa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Karin Dieperink nurse, MCN, Ph.d. student, Department of oncology Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S-20090142
Record Dates: First submitted 2011-01-05; First posted 2011-01-10 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2011-01

CONDITIONS: Urinary Irritative/Incontinence Problems; Bowel Problems; Sexual Problems; Hormonal Problems; Phycological Problems
Keywords: Rehabilitation; Coping; Prostate cancer; Nursing; Physiotherapy; Pelvic floor exercises; Motivational Interviewing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation (Active Comparator): note intervention
  Interventions: Behavioral: RePCa A
- Control (Placebo Comparator): same radiotherapy but no rehabilitation
  Interventions: Behavioral: RePCa A

INTERVENTIONS:
Behavioral: RePCa A — Intervention patients receives two consultations with a specialist oncology nurse three and six month after ended radiotherapy. The focus are on what is important for the patients at the specific time. The patient can bring his spouse.
  Furthermore the patients have two physiotherapy consultations with guidance in pelvic floor exercises and an individual home-program of pelvic and functional training exercises

SUMMARY:
This project will test and evaluate a rehabilitation programme, which will empower the mens health and give them resources to face at new everyday life.

The project examines if a focused interdisciplinary intervention has influence of the patients generic and specified quality of life after curative radiotherapy due to prostate cancer.

The intervention contains nursing consultation with information about late side effects, an individual plan and counselling in toilet habits, smoking cessation, weight control and psychological problems after treatment. Furthermore the patients are having physiotherapy with pelvic floor examinations. The nurse can refer to other collaborators.

DETAILED DESCRIPTION:
More cancer patients are now being cured or living a long time with the disease. Prostate cancer (PCa) is one of the cancer diseases, where the treatment can give some late side effects and cause reduced life quality.

This project will as a part of a ph.d. study, test and evaluate a rehabilitation programme, which will empower the mens health and give them resources to face at new everyday life.

The project is consisted of a randomised controlled test of the intervention and qualitative evaluation.

More and more Danish men are diagnosed with PC, the incidence increased with 34 percent from 2005-2007. This is caused partly due to a change in the age in the society and due to earlier diagnostics. PCa is now the most known cancer occurring in men in Denmark.

If the disease has not yet been metastasized, it is possible to use radiotherapy often in combination with anti hormones. It is possible to cure the patient, íf his disease is discovered in time, but there are some late side effects bond to the treatment, and they have influence of the patients quality of life. These are: impotence, incontinence, problem with the bowels, anxiety and depression.

The project is as followed:

Rehabilitation: Examine if a focused interdisciplinary intervention has influence of the patients generic and specified quality of life after curative radiotherapy due to prostate cancer. The intervention contains nursing consultation with information about late side effects, an individual plan and counselling in toilet habits, smoking cessation, weight control and psychological problems after treatment. Furthermore the patients are having physiotherapy with pelvic floor examinations. The nurse can refer to other collaborators.

Methods: Prospective randomised controlled study. Material: 160 patients are included. 80 patients in the intervention group and 80 patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized og locally advanced prostate cancer treated with curative intended radiotherapy at Department of Oncology Odense University Hospital in the period of inclusion

Exclusion Criteria:

* Patients younger than 18
* Patients who cannot understand/read or speak danish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
HRQOL urinary irritative score | 12 month
  The expanded prostate cancer Index Composite (EPIC)irritative score

SECONDARY OUTCOMES:
EMG measurement of pelvic floor muscles | 12 month
  Strength of pelvic floor muscles measured with electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Olfred Hansen, Dr. med Phd, Principal Investigator — Department of Oncology Odense University Hospital
Locations (1):
- Department of Oncology Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Dieperink KB, Johansen C, Hansen S, Wagner L, Andersen KK, Minet LR, Hansen O. The effects of multidisciplinary rehabilitation: RePCa-a randomised study among primary prostate cancer patients. Br J Cancer. 2013 Dec 10;109(12):3005-13. doi: 10.1038/bjc.2013.679. Epub 2013 Oct 29. PMID 24169342